CLINICAL TRIAL: NCT00202878
Title: A Multicenter, Double-Blind, Randomized Study to Establish the Clinical Benefit and Safety of Vytorin (Ezetimibe/Simvastatin Tablet) vs Simvastatin Monotherapy in High-Risk Subjects Presenting With Acute Coronary Syndrome (IMProved Reduction of Outcomes: Vytorin Efficacy International Trial - IMPROVE IT)
Brief Title: IMPROVE-IT: Examining Outcomes in Subjects With Acute Coronary Syndrome: Vytorin (Ezetimibe/Simvastatin) vs Simvastatin (P04103)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04103; MK-0653A-080 (Other: Merck Study Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Myocardial Infarction
Keywords: hypercholesterolemia; myocardial infarction; cholesterol; randomized controlled trials; acute coronary syndrome; angina
MeSH Terms: conditions — Hypercholesterolemia; Myocardial Infarction; Acute Coronary Syndrome; Angina Pectoris | interventions — Ezetimibe, Simvastatin Drug Combination; Simvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ezetimibe/simvastatin (Experimental): One Ezetimibe 10 mg/simvastatin 40 mg combination tablet and two simvastatin 40 mg placebo tablets once per day.
  Interventions: Drug: ezetimibe/simvastatin; Drug: Placebo for simvastatin 40 mg
- simvastatin (Active Comparator): One simvastatin 40 mg tablet, one ezetimibe/simvastatin combination 10/40 placebo tablet and one simvastatin 40 mg placebo tablet once per day.
  Interventions: Drug: simvastatin; Drug: Placebo for simvastatin 40 mg; Drug: Placebo for ezetimibe 10 mg/simvastatin 40 mg combination

INTERVENTIONS:
Drug: ezetimibe/simvastatin — Ezetimibe/simvastatin 10/40 mg per day from randomization through the end of participation. As per the original protocol, if LDL-C response was inadequate, the dose of simvastatin in the VYTORIN arm or simvastatin arm, could be increased to 80 mg (Note: per June 2011 protocol amendment, criteria for continued use of 80 mg simvastatin were modified and new increases of simvastatin dose to 80 mg were stopped).
  Other Names: Vytorin; Inegy
  Arms: ezetimibe/simvastatin
Drug: simvastatin — Simvastatin 40 mg per day from randomization through the end of participation. As per the original protocol, if LDL-C response was inadequate, the dose of simvastatin in the VYTORIN arm or simvastatin arm, could be increased to 80 mg (Note: per June 2011 protocol amendment, criteria for continued use of 80 mg simvastatin were modified and new increases of simvastatin dose to 80 mg were stopped).
  Other Names: Zocor
  Arms: simvastatin
Drug: Placebo for simvastatin 40 mg — one or two tablets orally daily
Drug: Placebo for ezetimibe 10 mg/simvastatin 40 mg combination — one tablet orally daily.
  Arms: simvastatin

SUMMARY:
This is a randomized, active-control, double-blind study of subjects with stabilized high-risk acute coronary syndrome (ACS). The primary objective is to evaluate the clinical benefit of Ezetimibe/Simvastatin Combination 10/40 (single tablet, under the brand VYTORIN in the United States) compared with Simvastatin 40 mg. As per the original protocol, if low-density lipoprotein cholesterol (LDL-C) response was inadequate, the dose of simvastatin in the VYTORIN arm or simvastatin arm, could be increased to 80 mg (Note: per June 2011 protocol amendment, criteria for continued use of 80 mg simvastatin were modified and new increases of simvastatin dose to 80 mg were stopped). Clinical benefit will be defined as the reduction in the risk of the occurrence of the composite endpoint of cardiovascular (CV) death, major coronary events, and stroke.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable participants may be eligible to enroll within 10 days following hospital admission with high-risk acute coronary syndrome (either ST-elevation myocardial infarction [STEMI] or Non-STEMI or unstable angina)
* Participants not taking a statin must have an LDL-C of 125 mg/dl or less. Participants taking a statin must have an LDL-C of 100 mg/dl or less.

Exclusion Criteria:

* Pregnant or lactating woman, or intending to become pregnant
* Participant with active liver disease or persistent unexplained serum transaminase elevation
* History of alcohol or drug abuse
* History of sensitivity to statin or ezetimibe
* A participant for whom discontinuation of existing lipid lowering regimen poses an unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18144 (Actual)
Dates: Start 2005-10-17 (Actual); Primary Completion 2014-09-18 (Actual); Study Completion 2014-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blazing MA, Giugliano RP, Cannon CP, Musliner TA, Tershakovec AM, White JA, Reist C, McCagg A, Braunwald E, Califf RM. Evaluating cardiovascular event reduction with ezetimibe as an adjunct to simvastatin in 18,144 patients after acute coronary syndromes: final baseline characteristics of the IMPROVE-IT study population. Am Heart J. 2014 Aug;168(2):205-12.e1. doi: 10.1016/j.ahj.2014.05.004. Epub 2014 May 15. PMID 25066560
- [Background] Califf RM, Lokhnygina Y, Cannon CP, Stepanavage ME, McCabe CH, Musliner TA, Pasternak RC, Blazing MA, Giugliano RP, Harrington RA, Braunwald E. An update on the IMProved reduction of outcomes: Vytorin Efficacy International Trial (IMPROVE-IT) design. Am Heart J. 2010 May;159(5):705-9. doi: 10.1016/j.ahj.2010.03.004. Epub 2010 Mar 15. No abstract available. PMID 20435175
- [Background] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Result] Bohula EA, Giugliano RP, Cannon CP, Zhou J, Murphy SA, White JA, Tershakovec AM, Blazing MA, Braunwald E. Achievement of dual low-density lipoprotein cholesterol and high-sensitivity C-reactive protein targets more frequent with the addition of ezetimibe to simvastatin and associated with better outcomes in IMPROVE-IT. Circulation. 2015 Sep 29;132(13):1224-33. doi: 10.1161/CIRCULATIONAHA.115.018381. Epub 2015 Sep 1. PMID 26330412
- [Derived] Cheng Y, Zhai S, Zhong W, West RM, Shen J. Improving polygenic risk score based drug response prediction using transfer learning. NPJ Genom Med. 2025 Nov 21;10(1):74. doi: 10.1038/s41525-025-00528-x. PMID 41271821
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Patel SM, Qamar A, Giugliano RP, Jarolim P, Marston NA, Park JG, Blazing MA, Cannon CP, Braunwald E, Morrow DA. Association of Serial High-Sensitivity Cardiac Troponin T With Subsequent Cardiovascular Events in Patients Stabilized After Acute Coronary Syndrome: A Secondary Analysis From IMPROVE-IT. JAMA Cardiol. 2022 Dec 1;7(12):1199-1206. doi: 10.1001/jamacardio.2022.3627. PMID 36260325
- [Derived] Fordyce CB, Giugliano RP, Cannon CP, Roe MT, Sharma A, Page C, White JA, Lokhnygina Y, Braunwald E, Blazing MA. Cardiovascular Events and Long-Term Risk of Sudden Death Among Stabilized Patients After Acute Coronary Syndrome: Insights From IMPROVE-IT. J Am Heart Assoc. 2022 Feb 15;11(4):e022733. doi: 10.1161/JAHA.121.022733. Epub 2022 Feb 3. PMID 35112882
- [Derived] Oyama K, Giugliano RP, Blazing MA, Park JG, Tershakovec AM, Sabatine MS, Cannon CP, Braunwald E. Baseline Low-Density Lipoprotein Cholesterol and Clinical Outcomes of Combining Ezetimibe With Statin Therapy in IMPROVE-IT. J Am Coll Cardiol. 2021 Oct 12;78(15):1499-1507. doi: 10.1016/j.jacc.2021.08.011. PMID 34620406
- [Derived] Giugliano RP, Gencer B, Wiviott SD, Park JG, Fuchs CS, Goessling W, Musliner TA, Tershakovec AM, Blazing MA, Califf R, Cannon CP, Braunwald E. Prospective Evaluation of Malignancy in 17,708 Patients Randomized to Ezetimibe Versus Placebo: Analysis From IMPROVE-IT. JACC CardioOncol. 2020 Sep 15;2(3):385-396. doi: 10.1016/j.jaccao.2020.07.008. eCollection 2020 Sep. PMID 34396246
- [Derived] Nanna MG, Navar AM, Giugliano RP, White JA, Lokhnygina Y, Mitchel YB, Musliner TA, Cannon CP, Blazing MA. Muscle Complaints or Events in Patients Randomized to Simvastatin or Ezetimibe/Simvastatin. J Am Coll Cardiol. 2020 Feb 25;75(7):835-837. doi: 10.1016/j.jacc.2019.12.022. No abstract available. PMID 32081289
- [Derived] Bach RG, Cannon CP, Giugliano RP, White JA, Lokhnygina Y, Bohula EA, Califf RM, Braunwald E, Blazing MA. Effect of Simvastatin-Ezetimibe Compared With Simvastatin Monotherapy After Acute Coronary Syndrome Among Patients 75 Years or Older: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2019 Sep 1;4(9):846-854. doi: 10.1001/jamacardio.2019.2306. PMID 31314050
- [Derived] Sharma A, Sun JL, Lokhnygina Y, Roe MT, Ahmad T, Desai NR, Blazing MA. Patient Phenotypes, Cardiovascular Risk, and Ezetimibe Treatment in Patients After Acute Coronary Syndromes (from IMPROVE-IT). Am J Cardiol. 2019 Apr 15;123(8):1193-1201. doi: 10.1016/j.amjcard.2019.01.034. Epub 2019 Jan 25. PMID 30739657
- [Derived] Navar AM, Roe MT, White JA, Cannon CP, Lokhnygina Y, Newby LK, Giugliano RP, Tershakovec AM, Braunwald E, Califf RM, Blazing MA. Medication Discontinuation in the IMPROVE-IT Trial. Circ Cardiovasc Qual Outcomes. 2019 Jan;12(1):e005041. doi: 10.1161/CIRCOUTCOMES.118.005041. PMID 30630361
- [Derived] Bonaca MP, Gutierrez JA, Cannon C, Giugliano R, Blazing M, Park JG, White J, Tershakovec A, Braunwald E. Polyvascular disease, type 2 diabetes, and long-term vascular risk: a secondary analysis of the IMPROVE-IT trial. Lancet Diabetes Endocrinol. 2018 Dec;6(12):934-943. doi: 10.1016/S2213-8587(18)30290-0. Epub 2018 Nov 2. PMID 30396865
- [Derived] Simon TG, Corey KE, Cannon CP, Blazing M, Park JG, O'Donoghue ML, Chung RT, Giugliano RP. The nonalcoholic fatty liver disease (NAFLD) fibrosis score, cardiovascular risk stratification and a strategy for secondary prevention with ezetimibe. Int J Cardiol. 2018 Nov 1;270:245-252. doi: 10.1016/j.ijcard.2018.05.087. Epub 2018 May 26. PMID 29903515
- [Derived] Giugliano RP, Cannon CP, Blazing MA, Nicolau JC, Corbalan R, Spinar J, Park JG, White JA, Bohula EA, Braunwald E; IMPROVE-IT (Improved Reduction of Outcomes: Vytorin Efficacy International Trial) Investigators. Benefit of Adding Ezetimibe to Statin Therapy on Cardiovascular Outcomes and Safety in Patients With Versus Without Diabetes Mellitus: Results From IMPROVE-IT (Improved Reduction of Outcomes: Vytorin Efficacy International Trial). Circulation. 2018 Apr 10;137(15):1571-1582. doi: 10.1161/CIRCULATIONAHA.117.030950. Epub 2017 Dec 20. PMID 29263150
- [Derived] Kato ET, Cannon CP, Blazing MA, Bohula E, Guneri S, White JA, Murphy SA, Park JG, Braunwald E, Giugliano RP. Efficacy and Safety of Adding Ezetimibe to Statin Therapy Among Women and Men: Insight From IMPROVE-IT (Improved Reduction of Outcomes: Vytorin Efficacy International Trial). J Am Heart Assoc. 2017 Nov 18;6(11):e006901. doi: 10.1161/JAHA.117.006901. PMID 29151034
- [Derived] Bohula EA, Wiviott SD, Giugliano RP, Blazing MA, Park JG, Murphy SA, White JA, Mach F, Van de Werf F, Dalby AJ, White HD, Tershakovec AM, Cannon CP, Braunwald E. Prevention of Stroke with the Addition of Ezetimibe to Statin Therapy in Patients With Acute Coronary Syndrome in IMPROVE-IT (Improved Reduction of Outcomes: Vytorin Efficacy International Trial). Circulation. 2017 Dec 19;136(25):2440-2450. doi: 10.1161/CIRCULATIONAHA.117.029095. Epub 2017 Sep 30. PMID 28972004
- [Derived] Pokharel Y, Chinnakondepalli K, Vilain K, Wang K, Mark DB, Davies G, Blazing MA, Giugliano RP, Braunwald E, Cannon CP, Cohen DJ, Magnuson EA. Impact of Ezetimibe on the Rate of Cardiovascular-Related Hospitalizations and Associated Costs Among Patients With a Recent Acute Coronary Syndrome: Results From the IMPROVE-IT Trial (Improved Reduction of Outcomes: Vytorin Efficacy International Trial). Circ Cardiovasc Qual Outcomes. 2017 May;10(5):e003201. doi: 10.1161/CIRCOUTCOMES.116.003201. PMID 28506979
- [Derived] Giugliano RP, Wiviott SD, Blazing MA, De Ferrari GM, Park JG, Murphy SA, White JA, Tershakovec AM, Cannon CP, Braunwald E. Long-term Safety and Efficacy of Achieving Very Low Levels of Low-Density Lipoprotein Cholesterol : A Prespecified Analysis of the IMPROVE-IT Trial. JAMA Cardiol. 2017 May 1;2(5):547-555. doi: 10.1001/jamacardio.2017.0083. PMID 28291866
- [Derived] Bohula EA, Morrow DA, Giugliano RP, Blazing MA, He P, Park JG, Murphy SA, White JA, Kesaniemi YA, Pedersen TR, Brady AJ, Mitchel Y, Cannon CP, Braunwald E. Atherothrombotic Risk Stratification and Ezetimibe for Secondary Prevention. J Am Coll Cardiol. 2017 Feb 28;69(8):911-921. doi: 10.1016/j.jacc.2016.11.070. PMID 28231942
- [Derived] Murphy SA, Cannon CP, Blazing MA, Giugliano RP, White JA, Lokhnygina Y, Reist C, Im K, Bohula EA, Isaza D, Lopez-Sendon J, Dellborg M, Kher U, Tershakovec AM, Braunwald E. Reduction in Total Cardiovascular Events With Ezetimibe/Simvastatin Post-Acute Coronary Syndrome: The IMPROVE-IT Trial. J Am Coll Cardiol. 2016 Feb 2;67(4):353-361. doi: 10.1016/j.jacc.2015.10.077. PMID 26821621
- [Derived] Azar RR, Badaoui G, Sarkis A, Azar M, Aydanian H, Harb S, Achkouty G, Kassab R. Effect of ezetimibe/atorvastatin combination on oxidized low density lipoprotein cholesterol in patients with coronary artery disease or coronary artery disease equivalent. Am J Cardiol. 2010 Jul 15;106(2):193-7. doi: 10.1016/j.amjcard.2010.03.016. PMID 20599002
- [Derived] Cannon CP, Giugliano RP, Blazing MA, Harrington RA, Peterson JL, Sisk CM, Strony J, Musliner TA, McCabe CH, Veltri E, Braunwald E, Califf RM; IMPROVE-IT Investigators. Rationale and design of IMPROVE-IT (IMProved Reduction of Outcomes: Vytorin Efficacy International Trial): comparison of ezetimbe/simvastatin versus simvastatin monotherapy on cardiovascular outcomes in patients with acute coronary syndromes. Am Heart J. 2008 Nov;156(5):826-32. doi: 10.1016/j.ahj.2008.07.023. Epub 2008 Sep 2. PMID 19061694
- [Derived] Peto R, Emberson J, Landray M, Baigent C, Collins R, Clare R, Califf R. Analyses of cancer data from three ezetimibe trials. N Engl J Med. 2008 Sep 25;359(13):1357-66. doi: 10.1056/NEJMsa0806603. Epub 2008 Sep 2. PMID 18765432
- [Derived] Drazen JM, Jarcho JA, Morrissey S, Curfman GD. Cholesterol lowering and ezetimibe. N Engl J Med. 2008 Apr 3;358(14):1507-8. doi: 10.1056/NEJMe0801842. Epub 2008 Mar 30. No abstract available. PMID 18376001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult men and women presenting with non-ST segment elevation myocardial infarction (NSTEMI) , STEMI, or hospitalized, documented unstable angina (UA) whom a percutaneous coronary intervention (PCI) was planned as management for the qualifying acute coronary syndrome (ACS) event were eligible for entry into the trial.
Pre-assignment Details: Study continued until a minimum of 5,250 participants had a primary endpoint event and each participant was followed for a minimum of 2.5 years.
Period: Overall Study
Arm/Group | Ezetimibe/Simvastatin | Simvastatin
Started | 9067 | 9077
Completed | 6868 | 6860
Not Completed | 2199 | 2217
Not completed — Death | 964 | 968
Not completed — Only Vital Status Known | 357 | 356
Not completed — Lost to Follow-up | 44 | 49
Not completed — Site Closure | 39 | 36
Not completed — Withdrawal by Subject | 795 | 808

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe/Simvastatin | Simvastatin | Total
Number analyzed (Participants) | 9067 | 9077 | 18144
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.7) | 63.6 (9.8) | 63.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2225 | 2191 | 4416
  Male | 6842 | 6886 | 13728

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Cardiovascular Death, Major Coronary Event, or Non-fatal Stroke (Kaplan-Meier Estimate of Percentage of Participants Experiencing a Qualifying Event)
Description: The time (in months) from study start to the first occurrence of any of the following clinical outcomes was recorded: cardiovascular death, major coronary Event (non-fatal myocardial infarction [MI], documented unstable angina [UA] requiring hospitalization, or coronary revascularization with percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) ≥ 30 days after randomization), or non-fatal Stroke. A Clinical Endpoints Committee (CEC) reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who experienced cardiovascular death, major coronary event, or non-fatal stroke within 7 years from randomization.
Time Frame: Up to approximately 9 years
Population: All participants who were randomly assigned to a treatment arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ezetimibe/Simvastatin | Simvastatin
Number analyzed (Participants) | 9067 | 9077
Percentage of Participants | 32.72 [31.63 to 33.85] | 34.67 [33.56 to 35.81]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Simvastatin; Test type: Superiority or Other; p = 0.016, Cox proportional hazard model; Covariates of the stratification factors (EARLY ACS trial, chronic prescription lipid-lowering experience, and high-risk ACS diagnosis) and treatment; Hazard Ratio (HR) = 0.936, 95% CI 2-sided [0.887 to 0.988] — Model includes events from randomization to last study visit

2. Secondary Outcome: Time to First Occurrence of Death From Any Cause, Major Coronary Event, or Non-fatal Stroke (Kaplan-Meier Estimate of Percentage of Participants Experiencing a Qualifying Event)
Description: The time (in months) from study start to the first occurrence of any of the following clinical outcomes was recorded: death from any cause, major coronary event (non-fatal myocardial infarction, documented unstable angina requiring hospitalization, or coronary revascularization with percutaneous coronary intervention or coronary artery bypass grafting ≥ 30 days after randomization), or non-fatal stroke. A Clinical Endpoints Committee (CEC) reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who experienced death from any cause, major coronary event, or non-fatal stroke within 7 years from randomization.
Time Frame: Up to approximately 9 years
Population: All participants who were randomly assigned to a treatment arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ezetimibe/Simvastatin | Simvastatin
Number analyzed (Participants) | 9067 | 9077
Percentage of Participants | 38.65 [37.52 to 39.81] | 40.25 [39.11 to 41.41]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Simvastatin; Test type: Superiority or Other; p = 0.035, Cox proportional hazard model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.948, 95% CI 2-sided [0.903 to 0.996] — Model includes events from randomization to last study visit

3. Secondary Outcome: Time to First Occurrence of Coronary Heart Disease (CHD) Death, Non-fatal MI, or Urgent Coronary Revascularization With PCI or CABG ≥ 30 Days After Randomization (Kaplan-Meier Estimate of Percentage of Participants Experiencing a Qualifying Event)
Description: The time (in months) from study start to the first occurrence of any of the following clinical outcomes was recorded: CHD death, non-fatal MI, or urgent coronary revascularization with PCI or CABG ≥ 30 days after randomization. A Clinical Endpoints Committee (CEC) reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who experienced CHD death, non-fatal MI, or urgent coronary revascularization with PCI or CABG ≥ 30 days after randomization within 7 years from randomization.
Time Frame: Up to approximately 9 years
Population: All participants who were randomly assigned to a treatment arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ezetimibe/Simvastatin | Simvastatin
Number analyzed (Participants) | 9067 | 9077
Percentage of Participants | 17.52 [16.62 to 18.46] | 18.88 [17.96 to 19.83]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Simvastatin; Test type: Superiority or Other; p = 0.016, Cox proportional hazard model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.912, 95% CI 2-sided [0.847 to 0.983] — Model includes events from randomization to last study visit

4. Secondary Outcome: Time to First Occurrence of CV Death, Nonfatal MI, UA With Hospitalization, All Revascularization Occurring ≥30 Days After Randomization, and Non-fatal Stroke (Kaplan-Meier Estimate of Percentage of Participants Experiencing a Qualifying Event)
Description: The time (in months) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, non-fatal MI, documented UA that requires admission into a hospital, all revascularization (including non-coronary) occurring at least 30 days after randomization, and non-fatal stroke. A Clinical Endpoints Committee (CEC) reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, non-fatal MI, unstable angina with hospitalization, all revascularization occurring ≥ 30 days after randomization, and non-fatal stroke within 7 Years from randomization.
Time Frame: Up to approximately 9 years
Population: All participants who were randomly assigned to a treatment arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ezetimibe/Simvastatin | Simvastatin
Number analyzed (Participants) | 9067 | 9077
Percentage of Participants | 34.49 [33.38 to 35.63] | 36.20 [35.07 to 37.34]
Statistical Analysis 1: Comparison: Ezetimibe/Simvastatin vs Simvastatin; Test type: Superiority or Other; p = 0.035, Cox proportional hazard model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.945, 95% CI 2-sided [0.897 to 0.996] — Model includes events from randomization to last study visit

ADVERSE EVENTS:
Time Frame: up to 30 days after last dose of study drug (Up to approximately 9 years maximum)
Description: Safety Population included all participants randomly assigned to a treatment arm.
Groups:
- Ezetimide/Simvastatin: One Ezetimibe 10 mg/simvastatin 40 mg combination tablet and two simvastatin 40 mg placebo tablets once per day.
Arm/Group | Ezetimide/Simvastatin | Simvastatin
Serious Adverse Events (participants affected / at risk) | 3640/9067 | 3649/9077
Other Adverse Events (participants affected / at risk) | 5486/9067 | 5472/9077
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimide/Simvastatin (N=9067) | Simvastatin (N=9077)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 71 (71) | 55 (55)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hilar Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypereosinophilic Syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphoid Tissue Hyperplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Retroperitoneal Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic Lesion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Systemic Mastocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Adams-Stokes Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 7 (7) | 4 (4)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Arrhythmia Supraventricular (Cardiac disorders) | 1 (1) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 140 (140) | 150 (150)
Atrial Flutter (Cardiac disorders) | 24 (24) | 28 (28)
Atrial Tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Atrial Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block (Cardiac disorders) | 11 (11) | 7 (7)
Atrioventricular Block Complete (Cardiac disorders) | 13 (13) | 9 (9)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular Block Second Degree (Cardiac disorders) | 5 (5) | 8 (8)
Atrioventricular Dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 27 (27) | 30 (30)
Bundle Branch Block (Cardiac disorders) | 1 (1) | 0 (0)
Bundle Branch Block Left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Aneurysm (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 5 (5) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac Pseudoaneurysm (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 2 (2) | 5 (5)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 5 (5) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 2 (2)
Cardiorenal Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Chronotropic Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Conduction Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Cor Pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Dissection (Cardiac disorders) | 0 (0) | 2 (2)
Coronary Artery Perforation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Dressler's Syndrome (Cardiac disorders) | 3 (3) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Heart Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 2 (2) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 (2) | 6 (6)
Left Ventricular Dysfunction (Cardiac disorders) | 4 (4) | 3 (3)
Mitral Valve Incompetence (Cardiac disorders) | 4 (4) | 8 (8)
Mitral Valve Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 9 (9) | 6 (6)
Pericardial Effusion (Cardiac disorders) | 10 (10) | 6 (6)
Pericardial Haemorrhage (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 14 (14) | 11 (11)
Pericarditis Constrictive (Cardiac disorders) | 0 (0) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 17 (17) | 19 (19)
Sinus Arrest (Cardiac disorders) | 2 (2) | 2 (2)
Sinus Arrhythmia (Cardiac disorders) | 4 (4) | 2 (2)
Sinus Bradycardia (Cardiac disorders) | 7 (7) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 16 (16) | 18 (18)
Tachycardia (Cardiac disorders) | 2 (2) | 6 (6)
Tachycardia Paroxysmal (Cardiac disorders) | 2 (2) | 0 (0)
Torsade De Pointes (Cardiac disorders) | 0 (0) | 1 (1)
Trifascicular Block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular Extrasystoles (Cardiac disorders) | 3 (3) | 6 (6)
Ventricular Fibrillation (Cardiac disorders) | 10 (10) | 8 (8)
Ventricular Tachycardia (Cardiac disorders) | 29 (29) | 42 (42)
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Adenomatous Polyposis Coli (Congenital, familial and genetic disorders) | 3 (3) | 0 (0)
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 3 (3) | 3 (3)
Bicuspid Aortic Valve (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital Spinal Cord Anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dermoid Cyst (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Epidermal Naevus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Foramen Magnum Stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 7 (7) | 4 (4)
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Multiple Lentigines Syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 2 (2) | 4 (4)
Sickle Cell Anaemia With Crisis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Deafness Neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness Unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Inner Ear Disorder (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Inner Ear Inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle Ear Effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 19 (19) | 25 (25)
Vertigo Positional (Ear and labyrinth disorders) | 5 (5) | 4 (4)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Adrenal Mass (Endocrine disorders) | 2 (2) | 2 (2)
Basedow's Disease (Endocrine disorders) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 5 (5) | 11 (11)
Hyperparathyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hyperparathyroidism Primary (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 5 (5)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 (1) | 1 (1)
Pituitary Haemorrhage (Endocrine disorders) | 0 (0) | 1 (1)
Postpartum Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid Cyst (Endocrine disorders) | 1 (1) | 1 (1)
Thyroid Disorder (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid Haemorrhage (Endocrine disorders) | 0 (0) | 1 (1)
Toxic Nodular Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Blindness Transient (Eye disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 15 (15) | 17 (17)
Cataract Nuclear (Eye disorders) | 3 (3) | 0 (0)
Corneal Scar (Eye disorders) | 1 (1) | 0 (0)
Diabetic Retinopathy (Eye disorders) | 5 (5) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Exfoliation Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Eye Disorder (Eye disorders) | 1 (1) | 3 (3)
Eye Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 2 (2)
Hyphaema (Eye disorders) | 1 (1) | 0 (0)
Lens Dislocation (Eye disorders) | 0 (0) | 2 (2)
Macular Degeneration (Eye disorders) | 1 (1) | 0 (0)
Macular Oedema (Eye disorders) | 0 (0) | 1 (1)
Optic Ischaemic Neuropathy (Eye disorders) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Retinal Artery Occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 4 (4) | 4 (4)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 3 (3) | 0 (0)
Vitreous Disorder (Eye disorders) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 3 (3) | 4 (4)
Abdominal Adhesions (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 15 (15) | 13 (13)
Abdominal Mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 41 (41) | 43 (43)
Abdominal Pain Lower (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 21 (21) | 14 (14)
Abdominal Wall Cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 4 (4) | 1 (1)
Anal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal Stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's Oesophagus (Gastrointestinal disorders) | 0 (0) | 6 (6)
Bezoar (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel Movement Irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac Disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 8 (8) | 13 (13)
Colitis Ischaemic (Gastrointestinal disorders) | 9 (9) | 12 (12)
Colitis Ulcerative (Gastrointestinal disorders) | 7 (7) | 5 (5)
Constipation (Gastrointestinal disorders) | 14 (14) | 15 (15)
Crohn's Disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cyclic Vomiting Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 15 (15)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticular Perforation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 11 (11) | 10 (10)
Diverticulum Intestinal (Gastrointestinal disorders) | 2 (2) | 6 (6)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diverticulum Oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal Polyp (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 7 (7) | 10 (10)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 3 (3) | 6 (6)
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Duodenogastric Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 11 (11) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 5 (5)
Enteritis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Enterocele (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epigastric Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Erosive Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Faecal Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Femoral Hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Disorder (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric Haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastric Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Polyps (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastric Ulcer (Gastrointestinal disorders) | 12 (12) | 18 (18)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 4 (4) | 5 (5)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 29 (29) | 39 (39)
Gastritis Erosive (Gastrointestinal disorders) | 4 (4) | 6 (6)
Gastritis Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroduodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal Disorder (Gastrointestinal disorders) | 3 (3) | 3 (3)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 60 (60) | 64 (64)
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 27 (27) | 33 (33)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 6 (6) | 3 (3)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 8 (8) | 7 (7)
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial Eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 10 (10) | 9 (9)
Hypertrophic Anal Papilla (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 11 (11) | 11 (11)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Inguinal Hernia (Gastrointestinal disorders) | 69 (69) | 51 (51)
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 3 (3) | 1 (1)
Intestinal Dilatation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal Infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Intestinal Mass (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal Obstruction (Gastrointestinal disorders) | 15 (15) | 11 (11)
Intestinal Perforation (Gastrointestinal disorders) | 4 (4) | 6 (6)
Intestinal Polyp (Gastrointestinal disorders) | 2 (2) | 8 (8)
Intestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestinal Ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Large Intestine Perforation (Gastrointestinal disorders) | 4 (4) | 4 (4)
Large Intestine Polyp (Gastrointestinal disorders) | 40 (40) | 58 (58)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 16 (16) | 13 (13)
Lumbar Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 5 (5) | 0 (0)
Melaena (Gastrointestinal disorders) | 10 (10) | 3 (3)
Mesenteric Artery Embolism (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric Artery Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (8) | 11 (11)
Oedematous Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Achalasia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Motility Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Spasm (Gastrointestinal disorders) | 3 (3) | 1 (1)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Oesophageal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 7 (7) | 9 (9)
Oral Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic Cyst (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pancreatic Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic Mass (Gastrointestinal disorders) | 2 (2) | 3 (3)
Pancreatic Pseudocyst (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 35 (35) | 28 (28)
Pancreatitis Acute (Gastrointestinal disorders) | 13 (13) | 17 (17)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Relapsing (Gastrointestinal disorders) | 2 (2) | 0 (0)
Parotid Gland Enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic Ulcer (Gastrointestinal disorders) | 2 (2) | 4 (4)
Peritoneal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngo-Oesophageal Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 15 (15) | 17 (17)
Rectal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Polyp (Gastrointestinal disorders) | 17 (17) | 6 (6)
Rectal Prolapse (Gastrointestinal disorders) | 4 (4) | 0 (0)
Rectal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectourethral Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal Haematoma (Gastrointestinal disorders) | 4 (4) | 2 (2)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Salivary Gland Calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 13 (13) | 14 (14)
Splenic Artery Aneurysm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tongue Dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 6 (6) | 11 (11)
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 3 (3) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 26 (26) | 25 (25)
Volvulus (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 8 (8) | 5 (5)
Adverse Drug Reaction (General disorders) | 1 (1) | 1 (1)
Adverse Event (General disorders) | 1 (1) | 1 (1)
Adverse Reaction (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 14 (14) | 18 (18)
Brca2 Gene Mutation (General disorders) | 0 (0) | 1 (1)
Catheter Site Haemorrhage (General disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 7 (7) | 3 (3)
Chills (General disorders) | 1 (1) | 1 (1)
Complication Of Device Insertion (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 3 (3) | 2 (2)
Cyst Rupture (General disorders) | 0 (0) | 1 (1)
Device Battery Issue (General disorders) | 0 (0) | 1 (1)
Device Breakage (General disorders) | 0 (0) | 1 (1)
Device Dislocation (General disorders) | 3 (3) | 1 (1)
Device Failure (General disorders) | 2 (2) | 0 (0)
Device Issue (General disorders) | 0 (0) | 1 (1)
Device Lead Damage (General disorders) | 1 (1) | 1 (1)
Device Lead Issue (General disorders) | 1 (1) | 1 (1)
Device Malfunction (General disorders) | 5 (5) | 3 (3)
Device Occlusion (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 3 (3)
Drug Withdrawal Syndrome (General disorders) | 1 (1) | 0 (0)
Fat Necrosis (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 9 (9) | 2 (2)
Feeling Cold (General disorders) | 1 (1) | 0 (0)
Feeling Hot (General disorders) | 0 (0) | 1 (1)
Fibrosis (General disorders) | 1 (1) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 1 (1)
General Physical Health Deterioration (General disorders) | 2 (2) | 2 (2)
Generalised Oedema (General disorders) | 1 (1) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 7 (7) | 7 (7)
Hernia Obstructive (General disorders) | 1 (1) | 0 (0)
Hyperplasia (General disorders) | 0 (0) | 2 (2)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 1 (1) | 1 (1)
Implant Site Extravasation (General disorders) | 0 (0) | 1 (1)
Implant Site Haematoma (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 1 (1)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0)
Injection Site Thrombosis (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 8 (8) | 8 (8)
Medical Device Complication (General disorders) | 3 (3) | 0 (0)
Metaplasia (General disorders) | 1 (1) | 1 (1)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 2 (2) | 0 (0)
Necrosis (General disorders) | 0 (0) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 14 (14) | 16 (16)
Oedema Peripheral (General disorders) | 4 (4) | 5 (5)
Pacemaker Generated Arrhythmia (General disorders) | 1 (1) | 0 (0)
Pacemaker Syndrome (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (4) | 1 (1)
Pelvic Mass (General disorders) | 1 (1) | 0 (0)
Polyp (General disorders) | 2 (2) | 2 (2)
Puncture Site Haemorrhage (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 24 (24) | 14 (14)
Stent-Graft Endoleak (General disorders) | 0 (0) | 1 (1)
Submandibular Mass (General disorders) | 1 (1) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 0 (0) | 5 (5)
Thrombosis In Device (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 3 (3) | 3 (3)
Ulcer Haemorrhage (General disorders) | 1 (1) | 1 (1)
Xerosis (General disorders) | 1 (1) | 0 (0)
Alcoholic Liver Disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile Duct Stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 7 (7) | 6 (6)
Biliary Colic (Hepatobiliary disorders) | 4 (4) | 2 (2)
Biliary Dyskinesia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Biliary Tract Disorder (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 4 (4) | 6 (6)
Cholangitis Acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 47 (47) | 73 (73)
Cholecystitis Acute (Hepatobiliary disorders) | 27 (27) | 26 (26)
Cholecystitis Chronic (Hepatobiliary disorders) | 3 (3) | 8 (8)
Cholelithiasis (Hepatobiliary disorders) | 78 (78) | 71 (71)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Cholesterolosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Disorder (Hepatobiliary disorders) | 5 (5) | 6 (6)
Gallbladder Pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder Perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder Polyp (Hepatobiliary disorders) | 1 (1) | 2 (2)
Granulomatous Liver Disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic Cirrhosis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Hepatic Cyst (Hepatobiliary disorders) | 6 (6) | 5 (5)
Hepatic Failure (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic Mass (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Hepatorenal Syndrome (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic Hepatitis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 2 (2) | 2 (2)
Liver Disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal Hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Allergy To Arthropod Sting (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 3 (3) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Autoimmune Disorder (Immune system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 2 (2) | 2 (2)
Hypersensitivity (Immune system disorders) | 8 (8) | 6 (6)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 2 (2) | 4 (4)
Abdominal Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Abdominal Wall Abscess (Infections and infestations) | 1 (1) | 3 (3)
Abdominal Wall Infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 4 (4)
Abscess Intestinal (Infections and infestations) | 1 (1) | 0 (0)
Abscess Jaw (Infections and infestations) | 1 (1) | 1 (1)
Abscess Limb (Infections and infestations) | 5 (5) | 7 (7)
Abscess Neck (Infections and infestations) | 1 (1) | 1 (1)
Abscess Oral (Infections and infestations) | 0 (0) | 1 (1)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Alpha Haemolytic Streptococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 11 (11) | 3 (3)
Appendiceal Abscess (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 33 (33) | 18 (18)
Appendicitis Perforated (Infections and infestations) | 7 (7) | 2 (2)
Arthritis Bacterial (Infections and infestations) | 4 (4) | 3 (3)
Arthritis Infective (Infections and infestations) | 4 (4) | 1 (1)
Bacteraemia (Infections and infestations) | 5 (5) | 3 (3)
Bacterial Infection (Infections and infestations) | 2 (2) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Biliary Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Blister Infected (Infections and infestations) | 1 (1) | 0 (0)
Brain Abscess (Infections and infestations) | 1 (1) | 0 (0)
Breast Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 49 (49) | 43 (43)
Bronchitis Bacterial (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis Viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 17 (17) | 14 (14)
Campylobacter Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter Infection (Infections and infestations) | 1 (1) | 0 (0)
Candida Infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 49 (49) | 63 (63)
Cellulitis Of Male External Genital Organ (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 3 (3)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 12 (12) | 4 (4)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 1 (1)
Clostridium Difficile Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0)
Colonic Abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 8 (8) | 7 (7)
Dengue Fever (Infections and infestations) | 5 (5) | 2 (2)
Device Related Infection (Infections and infestations) | 2 (2) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 3 (3) | 2 (2)
Diabetic Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea Infectious (Infections and infestations) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 34 (34) | 37 (37)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Echinococciasis (Infections and infestations) | 1 (1) | 0 (0)
Emphysematous Cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 3 (3)
Encephalitis Viral (Infections and infestations) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 3 (3) | 4 (4)
Endocarditis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis Enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Epidemic Nephropathy (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 5 (5) | 2 (2)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 18 (18) | 14 (14)
Escherichia Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Extradural Abscess (Infections and infestations) | 1 (1) | 2 (2)
Febrile Infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal Infection (Infections and infestations) | 1 (1) | 1 (1)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 3 (3) | 7 (7)
Gastroenteritis (Infections and infestations) | 51 (51) | 44 (44)
Gastroenteritis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Salmonella (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 5 (5) | 11 (11)
Gastrointestinal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 2 (2) | 1 (1)
Gingival Abscess (Infections and infestations) | 1 (1) | 0 (0)
Graft Infection (Infections and infestations) | 1 (1) | 0 (0)
Groin Abscess (Infections and infestations) | 2 (2) | 2 (2)
Groin Infection (Infections and infestations) | 0 (0) | 1 (1)
H1n1 Influenza (Infections and infestations) | 0 (0) | 2 (2)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter Gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 2 (2)
Hepatitis C (Infections and infestations) | 1 (1) | 2 (2)
Herpes Simplex Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 6 (6) | 7 (7)
Hiv Infection (Infections and infestations) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 0 (0) | 2 (2)
Incision Site Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Incision Site Infection (Infections and infestations) | 0 (0) | 1 (1)
Incisional Hernia Gangrenous (Infections and infestations) | 1 (1) | 0 (0)
Infected Bites (Infections and infestations) | 0 (0) | 1 (1)
Infected Cyst (Infections and infestations) | 0 (0) | 1 (1)
Infected Dermal Cyst (Infections and infestations) | 0 (0) | 1 (1)
Infected Skin Ulcer (Infections and infestations) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 12 (12) | 12 (12)
Infectious Colitis (Infections and infestations) | 2 (2) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 7 (7) | 2 (2)
Influenza (Infections and infestations) | 5 (5) | 6 (6)
Intervertebral Discitis (Infections and infestations) | 1 (1) | 2 (2)
Joint Abscess (Infections and infestations) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 2 (2) | 2 (2)
Klebsiella Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 16 (16) | 9 (9)
Localised Infection (Infections and infestations) | 4 (4) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 10 (10) | 11 (11)
Lower Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1)
Lung Abscess (Infections and infestations) | 0 (0) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1) | 3 (3)
Lyme Disease (Infections and infestations) | 2 (2) | 3 (3)
Lymph Node Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 2 (2)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Aseptic (Infections and infestations) | 1 (1) | 1 (1)
Meningitis Viral (Infections and infestations) | 1 (1) | 3 (3)
Myelitis (Infections and infestations) | 0 (0) | 1 (1)
Myringitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Necrotising Fasciitis (Infections and infestations) | 1 (1) | 1 (1)
Oesophageal Candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 4 (4)
Osteomyelitis (Infections and infestations) | 4 (4) | 10 (10)
Osteomyelitis Chronic (Infections and infestations) | 1 (1) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 2 (2)
Otitis Media Chronic (Infections and infestations) | 0 (0) | 1 (1)
Pancreas Infection (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 2 (2) | 0 (0)
Perineal Abscess (Infections and infestations) | 0 (0) | 2 (2)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 4 (4)
Peritonitis Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar Abscess (Infections and infestations) | 1 (1) | 0 (0)
Periumbilical Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pilonidal Cyst (Infections and infestations) | 1 (1) | 1 (1)
Pneumococcal Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 255 (255) | 242 (242)
Pneumonia Bacterial (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia Chlamydial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Influenzal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Pneumococcal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia Pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 0 (0) | 2 (2)
Post Procedural Infection (Infections and infestations) | 3 (3) | 4 (4)
Postoperative Abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 8 (8) | 13 (13)
Proctitis Infectious (Infections and infestations) | 0 (0) | 1 (1)
Prostate Infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous Colitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas Infection (Infections and infestations) | 1 (1) | 0 (0)
Psoas Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 15 (15) | 9 (9)
Pyelonephritis Acute (Infections and infestations) | 4 (4) | 4 (4)
Pyomyositis (Infections and infestations) | 1 (1) | 0 (0)
Q Fever (Infections and infestations) | 1 (1) | 0 (0)
Rectal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal Abscess (Infections and infestations) | 1 (1) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 10 (10) | 12 (12)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Rotavirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Scrotal Abscess (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 37 (37) | 33 (33)
Sepsis Syndrome (Infections and infestations) | 2 (2) | 0 (0)
Septic Encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 12 (12) | 12 (12)
Serratia Infection (Infections and infestations) | 0 (0) | 1 (1)
Shunt Infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 5 (5)
Skin Infection (Infections and infestations) | 2 (2) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 5 (5) | 5 (5)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Sternitis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Subacute Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 4 (4) | 9 (9)
Sweat Gland Infection (Infections and infestations) | 0 (0) | 1 (1)
Tick-Borne Fever (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth Abscess (Infections and infestations) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 2 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 3 (3) | 4 (4)
Tuberculosis (Infections and infestations) | 2 (2) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 15 (15) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 77 (77) | 79 (79)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 19 (19) | 19 (19)
Vestibular Neuronitis (Infections and infestations) | 3 (3) | 2 (2)
Viral Infection (Infections and infestations) | 6 (6) | 7 (7)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Wound Abscess (Infections and infestations) | 1 (1) | 1 (1)
Wound Infection (Infections and infestations) | 5 (5) | 4 (4)
Wound Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic Stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 8 (8) | 10 (10)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bursa Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Chance Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Clavicle Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 12 (12)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Electric Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye Penetration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 11 (11) | 12 (12)
Fat Embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 10 (10) | 6 (6)
Femur Fracture (Injury, poisoning and procedural complications) | 19 (19) | 22 (22)
Fibula Fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Foot Fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foreign Body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Fractured Ischium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured Sacrum (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gastroenteritis Radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 11 (11) | 8 (8)
Heat Exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat Illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat Stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 28 (28) | 23 (23)
Humerus Fracture (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Incision Site Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Incisional Hernia, Obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inflammation Of Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Jaw Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 8 (8) | 9 (9)
Joint Injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Kidney Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Kidney Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Limb Crushing Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 6 (6) | 8 (8)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 7 (7) | 11 (11)
Meniscus Injury (Injury, poisoning and procedural complications) | 8 (8) | 5 (5)
Mouth Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Multiple Injuries (Injury, poisoning and procedural complications) | 2 (2) | 7 (7)
Muscle Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Near Drowning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Open Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 9 (9) | 4 (4)
Pancreatic Leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Pelvic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Peripheral Nerve Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Periprosthetic Osteolysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post Concussion Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Gastric Surgery Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Postmastectomy Lymphoedema Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis Fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Pulmonary Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation Proctitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Renal Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 18 (18) | 16 (16)
Road Traffic Accident (Injury, poisoning and procedural complications) | 15 (15) | 8 (8)
Scapula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scrotal Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Shunt Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Silicosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skeletal Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Snake Bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Spinal Column Injury (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Spinal Cord Injury Cauda Equina (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 4 (4) | 9 (9)
Splenic Rupture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Sternal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sternal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma Site Ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Tendon Rupture (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Tibia Fracture (Injury, poisoning and procedural complications) | 4 (4) | 8 (8)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Tracheostomy Malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ulna Fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Urinary Bladder Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 11 (11) | 10 (10)
Vascular Pseudoaneurysm Ruptured (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Wound Dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Wound Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 0 (0)
Anticoagulation Drug Level Below Therapeutic (Investigations) | 0 (0) | 1 (1)
Blood Creatine Increased (Investigations) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 4 (4) | 4 (4)
Blood Creatinine Increased (Investigations) | 2 (2) | 0 (0)
Blood Glucose Abnormal (Investigations) | 0 (0) | 2 (2)
Blood Glucose Increased (Investigations) | 2 (2) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Orthostatic Decreased (Investigations) | 1 (1) | 0 (0)
Blood Urine Present (Investigations) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 1 (1) | 0 (0)
Clostridium Test Positive (Investigations) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 2 (2) | 2 (2)
Ejection Fraction Decreased (Investigations) | 2 (2) | 2 (2)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram Repolarisation Abnormality (Investigations) | 1 (1) | 0 (0)
Endoscopy (Investigations) | 1 (1) | 0 (0)
Endoscopy Gastrointestinal (Investigations) | 0 (0) | 1 (1)
Gastrointestinal Examination (Investigations) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 2 (2)
Heart Rate Decreased (Investigations) | 1 (1) | 0 (0)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0)
Heart Rate Irregular (Investigations) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 3 (3) | 2 (2)
International Normalised Ratio Decreased (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Laboratory Test Abnormal (Investigations) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 4 (4) | 3 (3)
Occult Blood Positive (Investigations) | 2 (2) | 0 (0)
Precancerous Cells Present (Investigations) | 1 (1) | 0 (0)
Prostatic Specific Antigen Increased (Investigations) | 6 (6) | 3 (3)
Psychiatric Evaluation (Investigations) | 0 (0) | 1 (1)
Total Lung Capacity Decreased (Investigations) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 2 (2) | 3 (3)
Tumour Marker Increased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 3 (3) | 1 (1)
Weight Increased (Investigations) | 1 (1) | 1 (1)
Abnormal Loss Of Weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cholesterosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 34 (34) | 22 (22)
Diabetes Mellitus (Metabolism and nutrition disorders) | 22 (22) | 29 (29)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 14 (14) | 22 (22)
Diabetes With Hyperosmolarity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic Complication (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Failure To Thrive (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 4 (4) | 9 (9)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (15) | 11 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 16 (16) | 3 (3)
Hyperosmolar State (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 20 (20) | 17 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (10) | 9 (9)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Overweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 11 (11) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (25) | 23 (23)
Arthritis (Musculoskeletal and connective tissue disorders) | 32 (32) | 23 (23)
Arthritis Reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 36 (36) | 34 (34)
Bone Lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Chest Wall Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest Wall Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (9)
Diastasis Recti Abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Epiphysitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Extraskeletal Ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Fracture Malunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (8)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Intervertebral Disc Displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 28 (28) | 35 (35)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint Instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower Extremity Mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 19 (19) | 18 (18)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Monarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Morphoea (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 34 (34) | 21 (21)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 13 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (20) | 12 (12)
Myalgia Intercostal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myofascial Pain Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 175 (175) | 159 (159)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (9)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (9)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 12 (12) | 18 (18)
Rheumatic Fever (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8)
Rib Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 21 (21) | 16 (16)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft Tissue Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 22 (22) | 27 (27)
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (12) | 12 (12)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Synovial Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper Extremity Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Abdominal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acoustic Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acute Monocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 6 (6)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 10 (10)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 9 (9)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 11 (11)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Adrenal Gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Anal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Atypical Fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 5 (5)
B-Cell Lymphoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-Cell Small Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 140 (140) | 157 (157)
Basosquamous Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Anorectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Benign Duodenal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Ear Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7)
Benign Neoplasm Of Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign Neoplasm Of Conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Neoplasm Of Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Benign Neoplasm Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Benign Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Benign Small Intestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (32) | 41 (41)
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Bladder Cancer Stage 0, With Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17) | 23 (23)
Bladder Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 9 (9)
Bladder Transitional Cell Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder Transitional Cell Carcinoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Transitional Cell Carcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bone Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bone Giant Cell Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bone Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (32) | 22 (22)
Breast Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 5 (5)
Bronchioloalveolar Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burkitt's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Carcinoid Tumour Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cardiac Valve Fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central Nervous System Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Chronic Lymphocytic Leukaemia Stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (23) | 29 (29)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (32) | 28 (28)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Colon Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Colon Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cranial Nerve Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ear Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Endocrine Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Enteropathy-Associated T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Essential Thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Extradural Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extramammary Paget's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Eye Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fallopian Tube Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Gallbladder Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 8 (8)
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 20 (20)
Gastrooesophageal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Haemangioma Of Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma Of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Haemangioma Of Spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hairy Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 7 (7)
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatobiliary Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Huerthle Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypergammaglobulinaemia Benign Monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Immunoblastic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Inflammatory Carcinoma Of The Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Inflammatory Pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Intraductal Papillary Mucinous Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal Papillary-Mucinous Carcinoma Of Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Intraocular Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Large Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large Cell Lung Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large Intestine Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3)
Laryngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Leiomyosarcoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyosarcoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo Maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 14 (14)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lobular Breast Carcinoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 16 (16)
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung Adenocarcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 13 (13)
Lung Carcinoma Cell Type Unspecified Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung Carcinoma Cell Type Unspecified Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung Carcinoma Cell Type Unspecified Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 5 (5)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 65 (65) | 66 (66)
Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 8 (8)
Lymphoproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28 (28) | 26 (26)
Malignant Melanoma In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (9)
Malignant Melanoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Neoplasm Of Ampulla Of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Neoplasm Of Eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Neoplasm Of Pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant Neoplasm Of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant Urinary Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Mantle Cell Lymphoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Medullary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 10 (10)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 4 (4)
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesenteric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Mesothelioma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases To Adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 10 (10)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 6 (6)
Metastases To Gastrointestinal Tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 9 (9)
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6)
Metastases To Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Metastases To Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases To Pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases To The Mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Metastatic Carcinoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Carcinoma Of The Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic Choriocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6)
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Monoclonal Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Mucoepidermoid Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mycosis Fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mycosis Fungoides Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Nasal Sinus Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Natural Killer-Cell Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Neoplasm Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 13 (13)
Non-Hodgkin's Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Non-Secretory Adenoma Of Pituitary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 8 (8)
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Non-Small Cell Lung Cancer Stage Iiia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ocular Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 8 (8)
Oesophageal Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oral Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17) | 20 (20)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Pancreatic Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Pelvic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pharyngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Pituitary Tumour Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 10 (10)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pleomorphic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pleomorphic Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleural Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pleural Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Prolactin-Producing Pituitary Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 123 (123) | 117 (117)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 7 (7)
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Prostate Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 11 (11)
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 7 (7)
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Renal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 11 (11)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 19 (19)
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Salivary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Salivary Gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Sarcomatoid Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18) | 12 (12)
Skin Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Small Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 7 (7)
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spindle Cell Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 84 (84) | 91 (91)
Squamous Cell Carcinoma Of Head And Neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 4 (4)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 11 (11)
Squamous Cell Carcinoma Of The Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of The Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Sweat Gland Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Thymoma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thymoma Malignant Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Thyroid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 9 (9)
Tongue Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tracheal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tracheal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 8 (8)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ureteral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ureteric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Ureteric Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary Bladder Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary Bladder Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 2 (2) | 1 (1)
Arachnoid Cyst (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic Nervous System Imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Balance Disorder (Nervous system disorders) | 2 (2) | 1 (1)
Brain Injury (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 9 (9) | 4 (4)
Carotid Sinus Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 3 (3) | 2 (2)
Central Nervous System Lesion (Nervous system disorders) | 1 (1) | 2 (2)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Cervical Cord Compression (Nervous system disorders) | 1 (1) | 0 (0)
Cervical Myelopathy (Nervous system disorders) | 3 (3) | 4 (4)
Cervical Radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Cervicobrachial Syndrome (Nervous system disorders) | 1 (1) | 3 (3)
Cognitive Disorder (Nervous system disorders) | 2 (2) | 1 (1)
Complex Partial Seizures (Nervous system disorders) | 2 (2) | 1 (1)
Complicated Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 12 (12) | 10 (10)
Dementia (Nervous system disorders) | 5 (5) | 6 (6)
Dementia Alzheimer's Type (Nervous system disorders) | 2 (2) | 3 (3)
Demyelination (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic Coma (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic Hyperglycaemic Coma (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic Neuropathy (Nervous system disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 30 (30) | 30 (30)
Encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Epilepsy (Nervous system disorders) | 5 (5) | 6 (6)
Extrapyramidal Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 1 (1) | 2 (2)
Guillain-Barre Syndrome (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 11 (11) | 13 (13)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 3 (3)
Hypertensive Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intercostal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial Aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 6 (6) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 3 (3)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 2 (2) | 5 (5)
Migraine With Aura (Nervous system disorders) | 0 (0) | 1 (1)
Motor Neurone Disease (Nervous system disorders) | 1 (1) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 3 (3)
Muscle Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia Gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Nerve Compression (Nervous system disorders) | 1 (1) | 0 (0)
Nervous System Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 3 (3) | 4 (4)
Neurological Symptom (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Normal Pressure Hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0)
Occipital Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 3 (3)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 2 (2)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Partial Seizures (Nervous system disorders) | 1 (1) | 1 (1)
Perineurial Cyst (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Pneumocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Polyneuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Polyneuropathy Chronic (Nervous system disorders) | 0 (0) | 1 (1)
Post Polio Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 16 (16) | 20 (20)
Radial Nerve Palsy (Nervous system disorders) | 2 (2) | 0 (0)
Radicular Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 4 (4) | 3 (3)
Sciatica (Nervous system disorders) | 4 (4) | 9 (9)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 1 (1)
Spinal Cord Ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Spondylitic Myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Status Epilepticus (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 107 (107) | 96 (96)
Tarsal Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Tension Headache (Nervous system disorders) | 1 (1) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Transient Global Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive To Stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Vascular Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 (0) | 2 (2)
Viith Nerve Paralysis (Nervous system disorders) | 3 (3) | 3 (3)
Vith Nerve Paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Vith Nerve Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal Behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 2 (2) | 2 (2)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 2 (2) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 12 (12) | 12 (12)
Anxiety Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 3 (3) | 4 (4)
Bipolar I Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar Ii Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Burnout Syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1) | 2 (2)
Confusional State (Psychiatric disorders) | 9 (9) | 7 (7)
Conversion Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 3 (3) | 3 (3)
Delirium Tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 19 (19) | 17 (17)
Disorientation (Psychiatric disorders) | 0 (0) | 3 (3)
Generalised Anxiety Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 1 (1) | 4 (4)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Disorder Due To A General Medical Condition (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 10 (10) | 9 (9)
Neurosis (Psychiatric disorders) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 3 (3) | 4 (4)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 2 (2) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Somatisation Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Somatoform Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 3 (3)
Suicide Attempt (Psychiatric disorders) | 4 (4) | 2 (2)
Withdrawal Syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Prerenal Failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder Diverticulum (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder Mass (Renal and urinary disorders) | 0 (0) | 3 (3)
Bladder Neck Obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder Neck Sclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder Obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder Perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder Prolapse (Renal and urinary disorders) | 1 (1) | 3 (3)
Bladder Spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder Tamponade (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus Bladder (Renal and urinary disorders) | 4 (4) | 4 (4)
Calculus Ureteric (Renal and urinary disorders) | 16 (16) | 11 (11)
Calculus Urethral (Renal and urinary disorders) | 1 (1) | 2 (2)
Calculus Urinary (Renal and urinary disorders) | 6 (6) | 3 (3)
Crush Syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis Noninfective (Renal and urinary disorders) | 3 (3) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 27 (27) | 20 (20)
Hydronephrosis (Renal and urinary disorders) | 5 (5) | 7 (7)
Hypertonic Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotonic Urinary Bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 31 (31) | 35 (35)
Nephropathy (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic Syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive Uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Aneurysm (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal Colic (Renal and urinary disorders) | 7 (7) | 2 (2)
Renal Cyst (Renal and urinary disorders) | 19 (19) | 22 (22)
Renal Cyst Ruptured (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Embolism (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 38 (38) | 29 (29)
Renal Failure Acute (Renal and urinary disorders) | 51 (51) | 61 (61)
Renal Failure Chronic (Renal and urinary disorders) | 12 (12) | 6 (6)
Renal Haemorrhage (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal Hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal Infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Mass (Renal and urinary disorders) | 3 (3) | 4 (4)
Renal Tubular Necrosis (Renal and urinary disorders) | 2 (2) | 2 (2)
Stress Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureteric Dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric Obstruction (Renal and urinary disorders) | 0 (0) | 3 (3)
Ureteric Stenosis (Renal and urinary disorders) | 1 (1) | 3 (3)
Urethral Caruncle (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral Dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral Stenosis (Renal and urinary disorders) | 9 (9) | 10 (10)
Urge Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Bladder Polyp (Renal and urinary disorders) | 1 (1) | 4 (4)
Urinary Incontinence (Renal and urinary disorders) | 7 (7) | 7 (7)
Urinary Retention (Renal and urinary disorders) | 14 (14) | 27 (27)
Urinary Tract Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Obstruction (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 72 (72) | 72 (72)
Breast Disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Cervical Dysplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 5 (5) | 3 (3)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Endometrial Hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Ovarian Cyst (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Ovarian Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Prolapse (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Penile Vein Thrombosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penis Disorder (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Peyronie's Disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatic Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic Disorder (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatic Dysplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatic Obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 5 (5) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 6 (6) | 2 (2)
Rectoprostatic Fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal Haematocoele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine Inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Polyp (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Uterine Prolapse (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Uterovaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Vaginal Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 12 (12)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 17 (17)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 109 (109) | 105 (105)
Chronic Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 (47) | 56 (56)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Dyspnoea Paroxysmal Nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 16 (16)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Laryngeal Cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal Polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal Ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Lung Hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Nasal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal Septum Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Turbinate Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 24 (24)
Pleural Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 9 (9)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 46 (46) | 36 (36)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pulmonary Granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 22 (22)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 32 (32) | 22 (22)
Restrictive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (8)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal Cord Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal Cord Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Vocal Cord Leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 12 (12) | 18 (18)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Campbell De Morgan Spots (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (7)
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Excessive Granulation Tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Granuloma Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen Planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichenoid Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmoplantar Keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pityriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Punctate Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 14 (14)
Skin Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 8 (8) | 6 (6)
Solar Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cardiac Assistance Device User (Social circumstances) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Arthrodesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder Catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac Rehabilitation Therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Fascia Release (Surgical and medical procedures) | 0 (0) | 1 (1)
Finger Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Gastric Bypass (Surgical and medical procedures) | 2 (2) | 0 (0)
Gastrointestinal Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia Repair (Surgical and medical procedures) | 1 (1) | 2 (2)
Hip Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip Surgery (Surgical and medical procedures) | 8 (8) | 9 (9)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Ileostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Immunoglobulin Therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 3 (3) | 1 (1)
Incisional Hernia Repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Intraocular Lens Implant (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint Arthroplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Knee Arthroplasty (Surgical and medical procedures) | 2 (2) | 1 (1)
Knee Operation (Surgical and medical procedures) | 13 (13) | 8 (8)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Mitral Valve Repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal Septal Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Penile Prosthesis Insertion (Surgical and medical procedures) | 2 (2) | 0 (0)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
Preoperative Care (Surgical and medical procedures) | 1 (1) | 0 (0)
Prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Rehabilitation Therapy (Surgical and medical procedures) | 3 (3) | 5 (5)
Rotator Cuff Repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Shoulder Operation (Surgical and medical procedures) | 3 (3) | 0 (0)
Spinal Decompression (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 7 (7) | 5 (5)
Suture Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral Bladder Resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral Prostatectomy (Surgical and medical procedures) | 2 (2) | 1 (1)
Turbinectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Varicose Vein Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Vertebroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Accelerated Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Aneurysm (Vascular disorders) | 1 (1) | 3 (3)
Angiodysplasia (Vascular disorders) | 2 (2) | 2 (2)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 29 (29) | 40 (40)
Aortic Aneurysm Rupture (Vascular disorders) | 2 (2) | 2 (2)
Aortic Dilatation (Vascular disorders) | 1 (1) | 2 (2)
Aortic Disorder (Vascular disorders) | 1 (1) | 0 (0)
Aortic Dissection (Vascular disorders) | 5 (5) | 4 (4)
Aortic Rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 9 (9) | 5 (5)
Arterial Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0)
Arterial Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous Fistula (Vascular disorders) | 1 (1) | 0 (0)
Behcet's Syndrome (Vascular disorders) | 1 (1) | 0 (0)
Blood Pressure Fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Blood Pressure Inadequately Controlled (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 19 (19) | 33 (33)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Essential Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Extremity Necrosis (Vascular disorders) | 2 (2) | 0 (0)
Femoral Artery Aneurysm (Vascular disorders) | 3 (3) | 2 (2)
Femoral Artery Occlusion (Vascular disorders) | 0 (0) | 2 (2)
Granulomatosis With Polyangiitis (Vascular disorders) | 3 (3) | 0 (0)
Haematoma (Vascular disorders) | 12 (12) | 16 (16)
Haemorrhage (Vascular disorders) | 5 (5) | 5 (5)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 25 (25) | 27 (27)
Hypertensive Crisis (Vascular disorders) | 21 (21) | 22 (22)
Hypertensive Emergency (Vascular disorders) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 27 (27) | 16 (16)
Hypovolaemic Shock (Vascular disorders) | 3 (3) | 2 (2)
Iliac Artery Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Intermittent Claudication (Vascular disorders) | 6 (6) | 6 (6)
Intra-Abdominal Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 3 (3) | 1 (1)
Jugular Vein Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Leriche Syndrome (Vascular disorders) | 0 (0) | 1 (1)
Lymphatic Fistula (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Malignant Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Necrosis Ischaemic (Vascular disorders) | 1 (1) | 0 (0)
Neurogenic Shock (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic Hypotension (Vascular disorders) | 10 (10) | 14 (14)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 5 (5) | 5 (5)
Peripheral Artery Aneurysm (Vascular disorders) | 4 (4) | 5 (5)
Peripheral Artery Stenosis (Vascular disorders) | 1 (1) | 3 (3)
Peripheral Artery Thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Peripheral Embolism (Vascular disorders) | 5 (5) | 7 (7)
Peripheral Ischaemia (Vascular disorders) | 2 (2) | 2 (2)
Peripheral Vascular Disorder (Vascular disorders) | 5 (5) | 4 (4)
Phlebitis (Vascular disorders) | 0 (0) | 3 (3)
Post Thrombotic Syndrome (Vascular disorders) | 1 (1) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Subclavian Artery Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Superior Vena Cava Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Superior Vena Cava Syndrome (Vascular disorders) | 0 (0) | 1 (1)
Temporal Arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 3 (3) | 3 (3)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Varicose Ulceration (Vascular disorders) | 0 (0) | 1 (1)
Varicose Vein (Vascular disorders) | 4 (4) | 5 (5)
Vascular Occlusion (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 1 (1)
Vasculitis Necrotising (Vascular disorders) | 0 (0) | 1 (1)
Venous Insufficiency (Vascular disorders) | 1 (1) | 3 (3)
Venous Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Venous Thrombosis Limb (Vascular disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimide/Simvastatin (N=9067) | Simvastatin (N=9077)
Diarrhoea (Gastrointestinal disorders) | 540 (540) | 552 (552)
Chest Pain (General disorders) | 694 (694) | 731 (731)
Fatigue (General disorders) | 720 (720) | 756 (756)
Non-Cardiac Chest Pain (General disorders) | 554 (554) | 543 (543)
Oedema Peripheral (General disorders) | 520 (520) | 551 (551)
Bronchitis (Infections and infestations) | 477 (477) | 450 (450)
Influenza (Infections and infestations) | 461 (461) | 483 (483)
Nasopharyngitis (Infections and infestations) | 618 (618) | 577 (577)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1001 (1001) | 914 (914)
Back Pain (Musculoskeletal and connective tissue disorders) | 866 (866) | 825 (825)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 616 (616) | 576 (576)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 581 (581) | 535 (535)
Myalgia (Musculoskeletal and connective tissue disorders) | 954 (954) | 908 (908)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 955 (955) | 899 (899)
Dizziness (Nervous system disorders) | 875 (875) | 909 (909)
Headache (Nervous system disorders) | 467 (467) | 520 (520)
Cough (Respiratory, thoracic and mediastinal disorders) | 702 (702) | 740 (740)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 787 (787) | 815 (815)
Hypertension (Vascular disorders) | 580 (580) | 642 (642)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All draft publications (eg, original manuscripts and abstracts of data and information relating to the IMPROVE-IT clinical study) shall be submitted to the Publication Committee at least 45 days prior to submission to a journal or public presentation.